CLINICAL TRIAL: NCT04541329
Title: Predicting Inflammatory Skin Disease Response to IL-23 Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-29813
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — tildrakizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tildrakizumab treatment (Experimental)
  Interventions: Biological: Tildrakizumab

INTERVENTIONS:
Biological: Tildrakizumab — IL-23 inhibitor

SUMMARY:
This study examines the effect of IL-23 blockade with Tildrakizumab on the immune cells of psoriatic skin lesions.

DETAILED DESCRIPTION:
This is a one-arm, open-label study to examine the effect of Tildrakizumab. Tildrakizumab is a FDA-approved medication for the treatment of cutaneous psoriasis. This study will examine how Tildrakizumab affects immune cells within psoriatic skin lesions. Fifteen subjects with moderate to severe psoriasis will be enrolled. Biopsy samples will be collected and undergo molecular profiling to correlate profiles with and to predict Tildrakizumab treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age at clinic visit.
* Documentation of moderate-severe psoriasis or atypical psoriasis.
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Tuberculosis, active serious infection, active systemic malignancy,
* Received a systemic medication for psoriasis within 3 months of study screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Cho, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tildrakizumab Treatment
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tildrakizumab Treatment
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 37 [30 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — country
  Participants
    United States | 7
Psoriasis Area and Severity Index (PASI) Score [Mean (Standard Deviation); unit: units on a scale] — Psoriasis Area and Severity Index (PASI) is a measure of psoriasis severity. The maximum score is 72, minimum score is 0. The higher the number, the more severe the psoriasis is.
  units on a scale | 10.7 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area and Severity Index (PASI) Score
Description: Psoriasis Area and Severity Index (PASI) is a measure of psoriasis severity. The maximum score is 72, minimum score is 0. The higher the number, the more severe the psoriasis is.
Time Frame: baseline and 3 months
Population: treated patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab Treatment
Number analyzed (Participants) | 7
score on a scale | 3.9 (4.1)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Tildrakizumab Treatment
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT04541329/Prot_SAP_002.pdf